CLINICAL TRIAL: NCT01241604
Title: Evaluation of Software Enhancements to the Respironics BiPAP autoSV Device Compared to BiPAP S/T Device
Acronym: SV3-ST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sub par recruitment performance
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MR-0830-ASV3-ST-SS
Record Dates: First submitted 2009-06-02; First posted 2010-11-16 (Estimated); Results first posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-03

CONDITIONS: Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Respironics BiPAP S/T (Active Comparator): Control Arm using Respironics BiPAP S/T
  Interventions: Device: BiPAP S/T
- Respironics BiPAP Auto SV3 (Active Comparator): Treatment arm using Respironics BiPAP Auto SV3
  Interventions: Device: BiPAP Auto SV3

INTERVENTIONS:
Device: BiPAP S/T — Mechanical Non-invasive Ventilation
  Other Names: Respironics BiPAP S/T
  Arms: Respironics BiPAP S/T
Device: BiPAP Auto SV3 — Auto Servo Ventilation Device
  Other Names: Respironics BiPAP auto SV Advanced
  Arms: Respironics BiPAP Auto SV3

SUMMARY:
This study is being undertaken to collect data from Respironics, Inc's BiPAP autoSV3 and compare with data from Respironics, Inc's BiPAP S/T device, to confirm that the algorithms in the BiPAP autoSV3 device can safely and effectively treat participants experiencing Comp SAS no worse than the BiPAP S/T device. This will be determined using a comparative, randomized design with the participants blinded to the therapy. Additionally, attempts will be made to blind the central scorer(s) with respect to which device is in use.

DETAILED DESCRIPTION:
Primary Hypothesis and end-point:

The use of the BiPAP autoSV3 device in participants with Comp SAS will treat those participants no worse than when compared to the BiPAP S/T device with respect to:

* Apnea-Hypopnea Index (AHI)

Secondary Hypothesis and end-points:

The use of the BiPAP autoSV3 device in participants with Comp SAS will treat those participants no worse than the BiPAP S/T device, with respect to:

* Sleep Variables
* REM, NREM and Total Sleep Time (TST) Indices
* Apnea Hypopnea Index (AHI)
* Center Apnea Index(CAI)
* Obstructive Apnea Index (OAI)
* Mixed Apnea Index (MAI)
* Hypopnea Index (HI)
* Sleep Onset Latency (SOL)
* REM Onset Latency (ROL)
* Wake After Sleep Onset (WASO)
* Total Sleep Time (TST)
* Sleep Efficiency (SE %)
* Wake (W), Stages N1,N2,N3 (NREM), and REM (R) sleep (in minutes)
* Wake (W), Stages N1,N2,N3 (NREM), and REM (R) sleep (% TST)
* Arousal Index [total, AH-related, PLM-related, 'spontaneous']
* Nocturnal oxygenation (measured by continuous pulse oximetry during sleep study)
* AHI (REM, NREM and TST) using modified hypopnea rule.
* AHI (REM, NREM and TST) during epochs for which leak is determined to exist within acceptable limits

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80.
* Ability to provide consent.
* Documentation of medical stability by investigator.
* Currently using BiPAP S/T (At least 4 weeks on therapy).
* Participants who previously demonstrated Complex Sleep Apnea (CSA), with a central apnea index (CAI) ≥5 during Diagnosis study or on Positive Airway Pressure (PAP) titration.

Exclusion Criteria:

* Participants, who are acutely ill, medically complicated or who are medically unstable.
* Participants in whom PAP therapy is otherwise medically contraindicated.
* Participants who are unwilling to wear PAP.
* Participants who are currently prescribed oxygen therapy.
* Participants with previously diagnosed respiratory failure or respiratory insufficiency and who are known to have chronically elevated arterial carbon dioxide levels while awake (PaCO2 ≥ 45mmHg).
* Participants who have had surgery of the upper airway, nose, sinus, or middle ear within the previous 90 days.
* Participants with untreated, non-obstructive sleep apnea (OSA)/CSA sleep disorders, including but not limited to; insomnia, periodic limb movement syndrome, or restless legs syndrome Periodic Limb Movement (PLM) Arousal Index > 15).
* Participants who are unwilling to participate in the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brydon Grant, MD, Principal Investigator — Medical Director of Med One Medical
Locations (1):
- Med One Medical Sleep Laboratory, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from one site to evaluate software enhancements. The study enrolled patients in the spring of 2009.
Groups:
- Screening Population: All participants that signed consent are considered for the screening population.
- Respironics BiPAP S/T First, Then Respironics BiPAP Auto SV3: Mechanical Non-invasive Ventilation first and then Auto Servo Ventilation Device
- Respironics BiPAP Auto SV3 First, Then Respironics BiPAP S/T: Auto Servo Ventilation Device and then Mechanical Non-invasive Ventilation
Period: Screening Period
Arm/Group | Screening Population | Respironics BiPAP S/T First, Then Respironics BiPAP Auto SV3 | Respironics BiPAP Auto SV3 First, Then Respironics BiPAP S/T
Started | 11 | 0 | 0
Completed | 8 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Screen Failure | 3 | 0 | 0
Period: Study Period
Arm/Group | Screening Population | Respironics BiPAP S/T First, Then Respironics BiPAP Auto SV3 | Respironics BiPAP Auto SV3 First, Then Respironics BiPAP S/T
Started | 0 | 5 | 3
Completed | 0 | 5 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The patients that were found eligible and were randomized are included in the baseline analysis.
Groups:
- All Participants: All participants that were consented.
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 8
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.8 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index
Description: The number of apneas and hypopneas per hour of sleep.
Time Frame: 2 nights
Population: One subject was excluded from analysis due to the subject chewing during the treatments causing the data to be unreliable.
  One subject had no pain related medical history and therefore was excluded from analysis.
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
events per hour | 19.24 (16.72) | 15.85 (17.24)
Statistical Analysis 1: Comparison: Respironics BiPAP S/T vs Respironics BiPAP Auto SV3; Test type: Equivalence — Equivalent non-parametric tests; p = .753, Wilcoxon signed ranks test

2. Secondary Outcome: Apnea Hypopnea Index- REM
Description: The apnea hypopneas index is the number of apneas and hypopneas per hour of sleep while in REM (Rapid eye movement sleep).
Time Frame: 2 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
events per hour | 10.16 (5.14) | 4.21 (4.49)

3. Secondary Outcome: Central Apnea Index
Description: The central apnea index is the number of central apneas divided by the number of hours of sleep.
Time Frame: 2 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
events per hour | 0.14 (0.25) | 0.11 (0.14)

4. Secondary Outcome: Obstructive Apnea Index
Description: The obstructive apnea index is the number of obstructive apneas per hour of sleep.
Time Frame: 2 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
events per hour | 0 (0) | 0 (0)

5. Secondary Outcome: Mixed Apnea Index
Description: The mixed apnea index is a combination of both obstructive and central sleep apnea symptoms per hour.
Time Frame: 2 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
events per hour | 0 (0) | 0 (0)

6. Secondary Outcome: Hypopnea Index
Description: The hypopnea index is number hypopneas per hour.
Time Frame: 2 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
events per hour | 19.1 (16.54) | 15.74 (17.23)

7. Secondary Outcome: Sleep Onset Latency
Description: Sleep Onset Latency is the amount of time it takes to fall asleep after the lights have been turned off.
Time Frame: 2 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
minutes | 43.25 (41.98) | 64.58 (81.64)

8. Secondary Outcome: REM Onset Latency
Description: REM Onset Latency is the time it takes to fall into REM sleep.
Time Frame: 2 nights
Population: This analysis was not done because this is not a standard measurement.
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Wake After Sleep Onset
Description: Wake After Sleep Onset is the amount time a participant is awake after they have fallen asleep.
Time Frame: 2 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
minutes | 72.58 (63.25) | 67.67 (39.86)

10. Secondary Outcome: Total Sleep Time
Description: Total Sleep time is total amount of time a participant is asleep from lights off to lights on.
Time Frame: 2 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
minutes | 331.83 (66.7) | 352.67 (63.5)

11. Secondary Outcome: Sleep Efficiency
Description: Sleep Efficiency is the percentage of time spent asleep while in bed.
Time Frame: 2 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time asleep
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
percentage of time asleep | 74.78 (12.36) | 73.42 (16.96)

12. Secondary Outcome: Periodic Limb Movement Index
Description: The periodic limb movement is the number of periodic limb movements per hour of sleep.
Time Frame: 2 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: movements per hour
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
movements per hour | 7.32 (10.4) | 4 (5.90)

13. Secondary Outcome: Arousal Index
Description: The arousal index is the number of arousals or awakenings per hour of sleep.
Time Frame: 2 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: arousals per hour
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
arousals per hour | 27.33 (14.3) | 23.76 (15.11)

14. Secondary Outcome: Stages N1,N2,N3 and REM (R) Sleep (% TST)
Description: The average amount of time spent N1, N2, N3 and REM percent total sleep time per night.
Time Frame: 2 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of TST per night
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
percentage of TST per night
  Stage N1 | 2.16 (2.95) | 1.37 (0.82)
  Stage N2 | 82.48 (15.54) | 83.44 (9.01)
  Stage N3 | 4.1 (8.14) | 4.27 (8.06)
  REM | 11.26 (8.13) | 10.92 (4.8)

15. Secondary Outcome: Stages N1,N2,N3 and REM (R) Sleep (in Minutes)
Description: The average amount of time spent N1, N2, N3 and REM in minutes per night.
Time Frame: 2 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
minutes
  Stage N1 | 7.17 (10.46) | 4.83 (3.33)
  Stage N2 | 271.33 (70.03) | 294.92 (67.18)
  Stage N3 | 15.25 (28.02) | 17.25 (23.01)
  REM | 37.92 (32.74) | 37.67 (17.44)

16. Secondary Outcome: Nocturnal Oxygenation Index
Description: Measurement of oxygen saturation index over the course of the night as measured by continuous pulse oximetry. The oxygen saturation index is the number of times per hour of sleep that the blood's oxygen level drop by a certain degree from baseline.
Time Frame: 2 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: oxygen saturation index
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 6 | 6
oxygen saturation index | 24 (24.9) | 19.93 (19.97)

17. Secondary Outcome: Apnea Hypopnea Index Using Modified Hypopnea Rule.
Description: The apnea hypopnea index is the number of apneas and hypopneas that occur per hour of sleep using the modified hypopnea rule.
Time Frame: 2 nights
Population: The Apnea Hyopnea Index(AHI) was analyzed and results were provided. The AHI using the modified hypopnea rule was not conducted. This is not part of the standard sleep scoring and therefore was not completed. The was an error in the endpoint analysis.
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Apnea Hypopnea Index(REM, NREM and TST) During Epochs for Which Leak is Determined to Exist Within Acceptable Limits.
Description: The number of apneas and hypopneas per hour of sleep during which the leak is determined to exist within acceptable limits.
Time Frame: 2 nights
Population: The Apnea Hypopnea Index (AHI) was analyzed and results were provided. However the epochs were not separated out as this is not part of the standard sleep scoring and therefore was not completed. The was an error in the endpoint analysis.
Arm/Group | Respironics BiPAP S/T | Respironics BiPAP Auto SV3
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 nights
Groups:
- Screening Period: All participants that were consented into the study.
- Respironics BiPAP Auto SV3 First, Then Respironics BiPAP S/T: Auto Servo Ventilation Device first and then Mechanical Non-invasive Ventilation
Arm/Group | Screening Period | Respironics BiPAP S/T First, Then Respironics BiPAP Auto SV3 | Respironics BiPAP Auto SV3 First, Then Respironics BiPAP S/T
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/11 | 0/5 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No